CLINICAL TRIAL: NCT03146845
Title: A Pilot Randomized Controlled Trial to Evaluate an Advanced Borderless Dressing (ALLEVYN LIFE Non-Bordered) in the Treatment of Chronic Ulcers
Brief Title: Evaluation Of An Advanced Borderless Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CT1603ALF
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2018-11

CONDITIONS: Pressure Ulcer; Leg Ulcer; Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Pressure Ulcer; Leg Ulcer
MeSH Terms: conditions — Pressure Ulcer; Leg Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ALLEVYN Life Non-Bordered (Experimental): Foam Dressing
  Interventions: Device: ALLEVYN Life Non-Bordered
- Standard care (Other): Standard care dressing
  Interventions: Device: Standard Care

INTERVENTIONS:
Device: ALLEVYN Life Non-Bordered — Foam Dressing
  Arms: ALLEVYN Life Non-Bordered
Device: Standard Care — Foam Dressing
  Arms: Standard care

SUMMARY:
This study will gather preliminary clinical, health economic, and safety data on the treatment of chronic wounds with the ALLEVYN Life Non-Bordered dressing compared to standard of care treatment when used on a wound.

DETAILED DESCRIPTION:
The study is a pilot RCT, which will generate the first comparative clinical, economic, and safety data for use of ALNB in subjects. A small sample of subjects with a range of chronic, moderate to highly exuding ulcer types (LU [arterial/mixed etiology leg ulcers or venous leg ulcers requiring compression therapy], PU, and non-ischemic DFU) will be enrolled and followed for 12 weeks to study the impact on health-related quality of life, ulcer progression and healthcare resource utilization.

ELIGIBILITY:
INCLUSION CRITERIA

1. The subject must provide informed consent to participate in the study.
2. The subject must be eighteen (18) years of age or older.
3. The subject must be willing and able to make all required study visits.
4. The subject must be able to follow instructions and be deemed capable of completing the CWIS questionnaire.
5. The subject must present with a chronic (≥ 4 weeks duration) ulcer which meets all of the following criteria:

   1. The ulcer is classified as either:

      * a pressure ulcer
      * a non-ischemic diabetic foot ulcer
      * a leg ulcer (arterial/mixed etiology leg ulcers or venous leg ulcers requiring compression therapy)
   2. The ulcer is, in the opinion of the Investigator, moderate to highly exuding.
   3. The ulcer would, in the opinion of the Investigator, benefit from a protective dressing.
   4. The ulcer is not infected based on clinical signs/symptoms.
6. A subject with a DFU must have an ankle-brachial index (ABI) of 0.7 or greater, as measured within 30 days of the Screening Visit.

EXCLUSION CRITERIA

1. Contraindications or hypersensitivity to the use of the ALLEVYN LIFE Non-Bordered, comparator, ancillary products, or their components.
2. Participation in the treatment period of another clinical trial within 30 days of Visit 1 or planned participation overlapping with this study.
3. The subject's reference ulcer is being treated with a topical antimicrobial dressing.
4. Subjects with skin features (e.g. tattoos, skin color, pre-existing scarring) which, in the opinion of the Investigator, could interfere with the study assessments.
5. Subjects who have participated previously in this clinical trial.
6. Subjects with a history of poor compliance with medical treatment.
7. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Winter, Study Director — Smith & Nephew, Inc.
Locations (6):
- United States (6):
  - Titan Clinical Solutions, Phoenix, Arizona
  - Center for Clinical Research, Martinez, California
  - UCLA Medical Center, Sylmar, California
  - Grace Research Ltd., Shreveport, Louisiana
  - Wound Care Plus, LLC, Summit, Missouri
  - JPS Health Network, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Started | 25 | 15
Completed | 20 | 11
Not Completed | 5 | 4
Not completed — Reference ulcer healed | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Noncompliance | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Surgeon applied a graft with non-removable dressing; discharged to surgeon's care | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care | Total
Number analyzed (Participants) | 25 | 15 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (15.5) | 53.7 (16.8) | 57.5 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 19 | 9 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 15 | 40
Height [Mean (Standard Deviation); unit: inches] | 67.9 (3.4) | 69.0 (4.1) | 68.3 (3.7)
Weight [Mean (Standard Deviation); unit: pounds] | 194.2 (65.6) | 230.5 (39.4) | 207.8 (59.3)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (9.4) | 34.1 (5.7) | 31.3 (8.4)
Reference Wound Type [Count of Participants; unit: Participants]
  Pressure ulcer | 5 | 2 | 7
  Diabetic foot ulcer | 12 | 8 | 20
  Venous leg ulcer | 8 | 4 | 12
  Mixed etiology ulcer | 0 | 1 | 1
  Other | 0 | 0 | 0
Wound Duration [Mean (Standard Deviation); unit: days] | 240.3 (166.6) | 292.9 (275.1) | 260.1 (211.9)
Wound Location [Count of Participants; unit: Participants]
  Head/neck | 0 | 0 | 0
  Shoulders | 0 | 0 | 0
  Upper arm | 0 | 0 | 0
  Lower arm | 0 | 0 | 0
  Wrist/hand | 0 | 0 | 0
  Chest | 0 | 0 | 0
  Abdomen | 0 | 0 | 0
  Back | 0 | 0 | 0
  Hips | 0 | 0 | 0
  Buttocks | 1 | 0 | 1
  Sacrum | 0 | 0 | 0
  Upper leg | 0 | 0 | 0
  Lower leg/knee | 5 | 4 | 9
  Ankle | 3 | 1 | 4
  Foot | 12 | 8 | 20
  Other | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in the Cardiff Wound Impact Schedule-Physical Symptoms of Daily Living (CWIS-PSDL) Scale Score From Baseline to the Week 6 Visit
Description: The primary objective was to estimate the effect of treatment with ALLEVYN Life Non-Bordered (ALNB) on Health-Related Quality of Life (HRQoL) in subjects with chronic ulcers, measured using the CWIS-PSDL scale, compared to subjects receiving standard care (SC) alone over a 6-week treatment period.
  The CWIS is a questionnaire to measure the impact of chronic wounds on patient health-related quality of life and identify areas of patient concern.
  The CWIS-PSDL score is transformed on to a 0-100 scale, where a high score indicates a positive rating. The following calculation is used:
  CWIS-PSDL = (Sum of PSDL item scores-N_PSDL)/(N_PSDL "x" 4) ×100, where NPSDL = count of 24 questions completed (experience and stress)
  PSDL Sub-scores are based on 24 questions (12 items on the extent of the problem and 12 on the associated stress), each graded on a 5-point Likert scale [1-5]) with higher scores indicating a better outcome.
Time Frame: Baseline through 6 weeks
Population: Scores were calculated for the full analysis set (FAS) population (all randomized subjects who received study treatment and attended at least 1 post-Baseline visit).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
score on a scale
  Baseline Assessment | 54.3 (27.5) | 54.0 (34.5)
  Week 6 Visit Assessment: number analyzed (Participants) | 24 | 13
  Week 6 Visit Assessment | 71.2 (24.4) | 56.3 (27.9)
  Change in CWIS-PSDL Scale Score: number analyzed (Participants) | 24 | 13
  Change in CWIS-PSDL Scale Score | 15.3 (23.3) | 2.3 (17.8)

2. Secondary Outcome: Change From Baseline CWIS-PSDL Score at 3 and 12 Weeks and CWIS-WB, CWIS-SL, CWIS-GQ, and CWIS-SQ Scores at 3, 6, and 12 Weeks
Description: Assessment of the change over time for the Cardiff Wound Impact Schedule-Physical Symptoms of Daily Living (CWIS-PSDL) Score at 3 and 12 weeks; CWIS-Well-Being (WB), CWIS-Social Life (SL), CWIS-Global Quality of Life (GQ), CWIS-Quality of Life Scales (SQ) at 3, 6, and 12 weeks.
  PSDL, SL, and WB sub-scores are based on 24 (score range 24-120), 14 (score range 14-70), and 7 (score range 7-35) questions, respectively; (each graded on a 5-point Likert scale [1-5])
  Higher scores on all CWIS metrics indicate a better outcome.
  PSDL score = (sum of PSDL item scores - 24)/96 x 100 = calculated score of 0 to 100; e.g., 95-24/96 x 100 = 74 (of a possible 100)
  WB Score = (sum of WB item scores - 7)/28 x 100 = calculated score of 0 to 100
  SL Score = (sum of SL item scores - 14)/56 x 100 = calculated score of 0 to 100
  GQ Score = "How good is your quality of life" = score range 0 to 10
  SQ Score = "How satisfied are you with your overall quality of life" = score range 0 to 10
Time Frame: PSDL: baseline, 3 and 12 weeks; WB, SL, GQ, and SQ: baseline, 3, 6, and 12 weeks
Population: Not all subjects participated in answering these questionnaire assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 24 | 13
score on a scale
  CWIS-PSDL Score Change at 3 Weeks | 6.0 (18.0) | 5.4 (35.6)
  CWIS-PSDL Score Change at 12 Weeks | 17.3 (22.1) | 16.6 (32.2)
  CWIS-WB Score Change at 3 Weeks | 9.5 (18.8) | 13.2 (25.7)
  CWIS-WB Score Change at 6 Weeks | 16.1 (23.1) | 4.9 (14.7)
  CWIS-WB Score Change at 12 Weeks | 19.2 (24.6) | 18.1 (28.5)
  CWIS-SL Score Change at 3 Weeks | 9.8 (22.9) | 8.1 (37.0)
  CWIS-SL Score Change at 6 Weeks | 14.9 (25.4) | 7.0 (26.7)
  CWIS-SL Score Change at 12 Weeks | 10.5 (32.4) | 16.1 (34.0)
  CWIS-GQ Change at 3 Weeks | -0.0 (3.1) | 0.8 (2.3)
  CWIS-GQ Change at 6 Weeks | 0.5 (2.5) | 0.7 (2.3)
  CWIS-GQ Change at 12 Weeks | 0.6 (2.3) | 1.1 (2.0)
  CWIS-SQ Change at 3 Weeks | 0.1 (3.2) | 1.1 (2.5)
  CWIS-SQ Change at 6 Weeks | 0.7 (2.5) | 1.1 (2.2)
  CWIS-SQ Change at 12 Weeks | 0.4 (2.3) | 0.8 (2.1)

3. Secondary Outcome: Ulcer Progression Using Modified Bates-Jensen Wound Assessment Tool (mBWAT) at Baseline, Weeks 3, 6, and 12 - Total Score
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) for an overall wound score at each time point.
  The mBWAT score combined the sub-scores of mBWAT - a tool that has been in widespread use since the early 1990s.
  mBWAT scoring: There are 13 categories of assessment with item-level score range of 1 to 5 on a modified Likert scale. Each item is scored for the wound characteristic it describes where 1 indicates least severe and 5 indicates most severe with higher scores indicating a more severe wound status. Scores taken over a period of time can be used to track the progression of the wound healing process. Possible score range from 13 to 65 for the total score.
  The 13 sub-categories include: Size, depth, edges, undermining, necrotic tissue type, necrotic tissue amount, exudate type, exudate amount, skin color surrounding wound, peripheral tissue edema, peripheral tissue induration, granulation tissue, and epithelialization
Time Frame: Baseline, Weeks 3, 6, and 12
Population: Not all subjects attended each scheduled visit and 2 subjects from the standard care group were withdrawn prior to receiving any treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
score on a scale
  Baseline Score | 19.8 (3.2) | 20 (4.2)
  Week 3 Score: number analyzed (Participants) | 23 | 11
  Week 3 Score | 18.5 (2.8) | 19.4 (4.4)
  Week 6 Score: number analyzed (Participants) | 23 | 11
  Week 6 Score | 17.3 (3.9) | 17.0 (2.9)
  Week 12 Score: number analyzed (Participants) | 23 | 11
  Week 12 Score | 16.4 (3.7) | 17.4 (5.7)

4. Secondary Outcome: Number of Participants With Each Type of Exudate; Analyzed for Ulcer Progression Using mBWAT - Individual Category Results
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) examining participants for the type of wound exudate exhibited at each time point.
  The tool defines the types of exudate as follows:
  Bloody = thin, bright red
  Serosanguinous = thin, watery, pale red to pink
  Serous = thin, watery, clear
  Purulent = thin or thick, opaque tan to yellow
  Foul purulent = thick, opaque yellow to green with offensive odor
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: None | 0 | 0
  Baseline: Bloody | 0 | 1
  Baseline: Serosanguineous | 12 | 7
  Baseline: Serous | 11 | 5
  Baseline: Purulent | 2 | 0
  Week 3: number analyzed (Participants) | 24 | 11
  Week 3: None | 1 | 0
  Week 3: Bloody | 0 | 0
  Week 3: Serosanguineous | 16 | 7
  Week 3: Serous | 6 | 4
  Week 3: Purulent | 1 | 0
  Week 6: number analyzed (Participants) | 24 | 11
  Week 6: None | 5 | 2
  Week 6: Bloody | 1 | 1
  Week 6: Serosanguineous | 9 | 3
  Week 6: Serous | 9 | 5
  Week 6: Purulent | 0 | 0
  Week 12: number analyzed (Participants) | 24 | 12
  Week 12: None | 11 | 5
  Week 12: Bloody | 2 | 1
  Week 12: Serosanguineous | 9 | 2
  Week 12: Serous | 2 | 3
  Week 12: Purulent | 0 | 1

5. Secondary Outcome: Number of Participants Per Category of Exudate Amount; Analyzed for Ulcer Progression Using mBWAT - Individual Category Results
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) examining participants for the amount of wound exudate demonstrated at each time point.
  The tool gives the following category descriptions for amount of exudate:
  None = wound tissues dry
  Scant = wound tissues moist; no measurable exudate
  Small = wound tissues wet; moisture evenly distributed in wound; drainage involves </=25% dressing
  Moderate = wound tissues saturated; drainage may or may not be evenly distributed in wound; drainage involves >25% to </=75% dressing
  Large = wound tissues bathed in fluid; drainage freely expressed; may or may not be evenly distributed in wound; drainage involves >75% dressing
  The tool advises to use a transparent metric measuring guide with concentric circles divided into 4 pie-shaped quadrants to determine percentage of dressing involved with exudate.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: None | 0 | 0
  Baseline: Scant, wound, moist but no observable exudate | 0 | 0
  Baseline: Small | 0 | 0
  Baseline: Moderate | 21 | 11
  Baseline: Large | 4 | 2
  Week 3: number analyzed (Participants) | 24 | 11
  Week 3: None | 1 | 0
  Week 3: Scant, wound, moist but no observable exudate | 1 | 1
  Week 3: Small | 11 | 3
  Week 3: Moderate | 7 | 5
  Week 3: Large | 4 | 2
  Week 6: number analyzed (Participants) | 24 | 11
  Week 6: None | 5 | 2
  Week 6: Scant, wound, moist but no observable exudate | 2 | 2
  Week 6: Small | 7 | 2
  Week 6: Moderate | 6 | 4
  Week 6: Large | 4 | 1
  Week 12: number analyzed (Participants) | 24 | 12
  Week 12: None | 11 | 5
  Week 12: Scant, wound, moist but no observable exudate | 1 | 1
  Week 12: Small | 6 | 1
  Week 12: Moderate | 3 | 4
  Week 12: Large | 3 | 1

6. Secondary Outcome: Number of Participants Per Category of Undermining; Analyzed for Ulcer Progression Using mBWAT - Individual Category Results
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) examining participants for the extent (measurement) of wound undermining at each time point.
  The tool guidance is as follows:
  Assess by inserting a cotton-tipped applicator under the wound edge;
  Advance it as far as it will go without using undue force;
  Raise the tip of the applicator so it may be seen or felt on the surface of the skin;
  Mark the surface with a pen;
  Measure the distance from the mark on the skin to the edge of the wound;
  Continue process around the wound;
  Then use a transparent metric measuring guide with concentric circles divided into 4 (25%) pie-shaped quadrants to help determine percent of wound involved.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: None present | 19 | 11
  Baseline: <2 cm in any area | 4 | 2
  Baseline: 2-4 cm involving <50% wound margins | 2 | 0
  Baseline: 2-4 cm involving >50% wound margins | 0 | 0
  Baseline: >4 cm or tunnelling in any area | 0 | 0
  Week 3: number analyzed (Participants) | 24 | 11
  Week 3: None present | 21 | 9
  Week 3: <2 cm in any area | 3 | 2
  Week 3: 2-4 cm involving <50% wound margins | 0 | 0
  Week 3: 2-4 cm involving >50% wound margins | 0 | 0
  Week 3: >4 cm or tunnelling in any area | 0 | 0
  Week 6: number analyzed (Participants) | 24 | 11
  Week 6: None present | 23 | 11
  Week 6: <2 cm in any area | 1 | 0
  Week 6: 2-4 cm involving <50% wound margins | 0 | 0
  Week 6: 2-4 cm involving >50% wound margins | 0 | 0
  Week 6: >4 cm or tunnelling in any area | 0 | 0
  Week 12: number analyzed (Participants) | 24 | 12
  Week 12: None present | 23 | 12
  Week 12: <2 cm in any area | 1 | 0
  Week 12: 2-4 cm involving <50% wound margins | 0 | 0
  Week 12: 2-4 cm involving >50% wound margins | 0 | 0
  Week 12: >4 cm or tunnelling in any area | 0 | 0

7. Secondary Outcome: Number of Participants Per Category of Type of Necrotic Tissue; Analyzed for Ulcer Progression Using mBWAT - Individual Category Results
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) examining participants for type (appearance) of necrotic tissue at each time point.
  The tool defines the categories of necrotic tissue type as follows:
  White/gray non-viable tissue = may appear prior to wound opening; skin surface is white or gray
  Non-adherent, yellow slough = thin, mucinous substance; scattered throughout wound bed; easily separated from wound tissue
  Loosely adherent, yellow slough = thick, stringy, clumps of debris; attached to wound tissue
  Adherent, soft, black eschar = soggy tissue; strongly attached to tissue in center or base of wound
  Firmly adherent, hard/black eschar = firm, crusty tissue; strongly attached to wound base and edges (like a hard scab)
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: None | 19 | 10
  Baseline: White/grey nonviable tissue and/or nonadherent yellow slough | 3 | 0
  Baseline: Loosely adherent yellow slough | 3 | 1
  Baseline: Adherent, soft, black eschar | 0 | 2
  Baseline: Firmly adherent, hard, black eschar | 0 | 0
  Week 3: number analyzed (Participants) | 23 | 11
  Week 3: None | 18 | 8
  Week 3: White/grey nonviable tissue and/or nonadherent yellow slough | 2 | 0
  Week 3: Loosely adherent yellow slough | 1 | 2
  Week 3: Adherent, soft, black eschar | 1 | 0
  Week 3: Firmly adherent, hard, black eschar | 1 | 1
  Week 6: number analyzed (Participants) | 23 | 11
  Week 6: None | 18 | 10
  Week 6: White/grey nonviable tissue and/or nonadherent yellow slough | 2 | 0
  Week 6: Loosely adherent yellow slough | 2 | 0
  Week 6: Adherent, soft, black eschar | 1 | 1
  Week 6: Firmly adherent, hard, black eschar | 0 | 0
  Week 12: number analyzed (Participants) | 23 | 11
  Week 12: None | 18 | 10
  Week 12: White/grey nonviable tissue and/or nonadherent yellow slough | 1 | 0
  Week 12: Loosely adherent yellow slough | 2 | 0
  Week 12: Adherent, soft, black eschar | 2 | 0
  Week 12: Firmly adherent, hard, black eschar | 0 | 1

8. Secondary Outcome: Number of Participants by the Amount of Necrotic Tissue Present; Analyzed for Ulcer Progression Using mBWAT - Individual Category Results
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) examining participants for the amount of necrotic tissue observed during dressing change at each time point.
  The tool guidance is to use a transparent metric measuring guide with concentric circles divided into 4 pie-shaped quadrants to help determine percent of wound involved.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: None | 19 | 10
  Baseline: <25% of wound bed covered | 4 | 1
  Baseline: 25% to 50% of wound covered | 1 | 1
  Baseline: >50% to <75% of wound covered | 0 | 0
  Baseline: >75% to 100% of wound covered | 1 | 1
  Week 3: number analyzed (Participants) | 23 | 11
  Week 3: None | 18 | 8
  Week 3: <25% of wound bed covered | 2 | 2
  Week 3: 25% to 50% of wound covered | 3 | 0
  Week 3: >50% to <75% of wound covered | 0 | 1
  Week 3: >75% to 100% of wound covered | 0 | 0
  Week 6: number analyzed (Participants) | 23 | 11
  Week 6: None | 18 | 10
  Week 6: <25% of wound bed covered | 4 | 0
  Week 6: 25% to 50% of wound covered | 1 | 1
  Week 6: >50% to <75% of wound covered | 0 | 0
  Week 6: >75% to 100% of wound covered | 0 | 0
  Week 12: number analyzed (Participants) | 23 | 11
  Week 12: None | 18 | 10
  Week 12: <25% of wound bed covered | 4 | 0
  Week 12: 25% to 50% of wound covered | 1 | 0
  Week 12: >50% to <75% of wound covered | 0 | 0
  Week 12: >75% to 100% of wound covered | 0 | 1

9. Secondary Outcome: Number of Participants With Skin Color Changes of the Surrounding Wound; Analyzed for Ulcer Progression Using mBWAT - Individual Category Results
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) examining participants for the appearance of skin color changes surrounding the reference wound at each time point.
  The tool guidance is to assess tissues within 4 cm of wound edge. Dark-skinned persons show the colors "bright red" and "dark red" as a deepening of normal ethnic skin color or a purple hue. As healing occurs in dark-skinned persons, the new skin is pink and may never darken.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: Pink or normal for ethnic group | 22 | 12
  Baseline: Bright red and/or blanches to touch | 3 | 0
  Baseline: White or grey pallor or hypopigmented | 0 | 0
  Baseline: Dark red/ or purple and/or nonblanchable | 0 | 1
  Baseline: Black or hyperpigmented | 0 | 0
  Week 3: number analyzed (Participants) | 23 | 11
  Week 3: Pink or normal for ethnic group | 23 | 10
  Week 3: Bright red and/or blanches to touch | 0 | 0
  Week 3: White or grey pallor or hypopigmented | 0 | 1
  Week 3: Dark red/ or purple and/or nonblanchable | 0 | 0
  Week 3: Black or hyperpigmented | 0 | 0
  Week 6: number analyzed (Participants) | 23 | 11
  Week 6: Pink or normal for ethnic group | 23 | 10
  Week 6: Bright red and/or blanches to touch | 0 | 1
  Week 6: White or grey pallor or hypopigmented | 0 | 0
  Week 6: Dark red/ or purple and/or nonblanchable | 0 | 0
  Week 6: Black or hyperpigmented | 0 | 0
  Week 12: number analyzed (Participants) | 23 | 11
  Week 12: Pink or normal for ethnic group | 23 | 9
  Week 12: Bright red and/or blanches to touch | 0 | 0
  Week 12: White or grey pallor or hypopigmented | 0 | 1
  Week 12: Dark red/ or purple and/or nonblanchable | 0 | 1
  Week 12: Black or hyperpigmented | 0 | 0

10. Secondary Outcome: Number of Participants With Granulation Tissue; Analyzed for Ulcer Progression Using mBWAT - Individual Category Results
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) examining participants for the appearance and percentage of granulation tissue in the reference wound at each time point.
  Granulation tissue is the growth of small blood vessels and connective tissue to fill in full-thickness wounds. Tissue is healthy when bright, beefy red, shiny, and granular with a velvety appearance. Poor vascular supply appears as pale-pink or blanched to dull, dusky red color.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: Skin intact or partial-thickness wound | 0 | 0
  Baseline: Bright, beefy red; 75-100% wound filled/ or tissue overgrowth | 10 | 6
  Baseline: Bright, beefy red; <75% & >25% wound filled | 8 | 2
  Baseline: Pink and/or dull, dusky red and/or fills ≤25% of wound | 7 | 4
  Baseline: No granulation tissue present | 0 | 1
  Week 3: number analyzed (Participants) | 23 | 11
  Week 3: Skin intact or partial-thickness wound | 0 | 0
  Week 3: Bright, beefy red; 75-100% wound filled/ or tissue overgrowth | 10 | 6
  Week 3: Bright, beefy red; <75% & >25% wound filled | 8 | 2
  Week 3: Pink and/or dull, dusky red and/or fills ≤25% of wound | 5 | 3
  Week 3: No granulation tissue present | 0 | 0
  Week 6: number analyzed (Participants) | 23 | 11
  Week 6: Skin intact or partial-thickness wound | 2 | 0
  Week 6: Bright, beefy red; 75-100% wound filled/ or tissue overgrowth | 9 | 8
  Week 6: Bright, beefy red; <75% & >25% wound filled | 9 | 3
  Week 6: Pink and/or dull, dusky red and/or fills ≤25% of wound | 3 | 0
  Week 6: No granulation tissue present | 0 | 0
  Week 12: number analyzed (Participants) | 23 | 11
  Week 12: Skin intact or partial-thickness wound | 2 | 0
  Week 12: Bright, beefy red; 75-100% wound filled/ or tissue overgrowth | 11 | 8
  Week 12: Bright, beefy red; <75% & >25% wound filled | 8 | 3
  Week 12: Pink and/or dull, dusky red and/or fills ≤25% of wound | 2 | 0
  Week 12: No granulation tissue present | 0 | 0

11. Secondary Outcome: Number of Participants With Epithelialization; Analyzed for Ulcer Progression Using mBWAT - Individual Category Results
Description: Assessment of ulcer progression by the modified Bates-Jensen Wound Assessment Tool (mBWAT) examining participants for the percentage of reference wound demonstrating epithelialization at each time point.
  Epithelialization is the process of epidermal resurfacing and appears as pink or red skin. In partial-thickness wounds, it can occur throughout the wound bed as well as from the wound edges. In full-thickness wounds, it occurs from the edges only.
  Use a transparent metric measuring guide with concentric circles divided into 4 (25%) pie-shaped quadrants to help determine percent of wound involved and to measure the distance the epithelial tissue extends into the wound.
  The mBWAT 13 categories include: Size, depth, edges, undermining, necrotic tissue type, necrotic tissue amount, exudate type, exudate amount, skin color surrounding wound, peripheral tissue edema, peripheral tissue induration, granulation tissue, and epithelialization.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: 100% wound covered, surface intact | 0 | 0
  Baseline: 75% - <100% wound covered and/or epithelial tissue extends >0.5 cm into wound bed | 6 | 4
  Baseline: 50% - <75% wound covered and/or epithelial tissue extends <0.5 cm into wound bed | 1 | 0
  Baseline: 25% - <50% wound covered | 5 | 1
  Baseline: <25% wound covered | 13 | 8
  Week 3: number analyzed (Participants) | 24 | 11
  Week 3: 100% wound covered, surface intact | 1 | 0
  Week 3: 75% - <100% wound covered and/or epithelial tissue extends >0.5 cm into wound bed | 6 | 3
  Week 3: 50% - <75% wound covered and/or epithelial tissue extends <0.5 cm into wound bed | 3 | 0
  Week 3: 25% - <50% wound covered | 4 | 2
  Week 3: <25% wound covered | 10 | 6
  Week 6: number analyzed (Participants) | 24 | 11
  Week 6: 100% wound covered, surface intact | 2 | 1
  Week 6: 75% - <100% wound covered and/or epithelial tissue extends >0.5 cm into wound bed | 6 | 2
  Week 6: 50% - <75% wound covered and/or epithelial tissue extends <0.5 cm into wound bed | 3 | 2
  Week 6: 25% - <50% wound covered | 2 | 2
  Week 6: <25% wound covered | 11 | 4
  Week 12: number analyzed (Participants) | 24 | 12
  Week 12: 100% wound covered, surface intact | 9 | 5
  Week 12: 75% - <100% wound covered and/or epithelial tissue extends >0.5 cm into wound bed | 5 | 4
  Week 12: 50% - <75% wound covered and/or epithelial tissue extends <0.5 cm into wound bed | 3 | 0
  Week 12: 25% - <50% wound covered | 3 | 1
  Week 12: <25% wound covered | 4 | 2

12. Secondary Outcome: Number of Participants With Peri-Wound Changes; Analyzed for Ulcer Progression Assessed by Condition
Description: Evaluation of the number of participants demonstrating peri-wound changes in appearance as determined visually by the Investigator; categorized as normal, erythematous, edematous, eczematous, excoriated, macerated, or indurated at each time point.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants
  Baseline: Normal | 22 | 11
  Baseline: Erythematous | 0 | 0
  Baseline: Edematous | 0 | 1
  Baseline: Eczematous | 1 | 1
  Baseline: Excoriated | 0 | 0
  Baseline: Macerated | 1 | 0
  Baseline: Indurated | 1 | 0
  Week 3: number analyzed (Participants) | 23 | 11
  Week 3: Normal | 20 | 9
  Week 3: Erythematous | 0 | 0
  Week 3: Edematous | 0 | 1
  Week 3: Eczematous | 1 | 1
  Week 3: Excoriated | 0 | 0
  Week 3: Macerated | 1 | 0
  Week 3: Indurated | 1 | 0
  Week 6: number analyzed (Participants) | 23 | 11
  Week 6: Normal | 20 | 8
  Week 6: Erythematous | 0 | 0
  Week 6: Edematous | 0 | 1
  Week 6: Eczematous | 0 | 1
  Week 6: Excoriated | 0 | 0
  Week 6: Macerated | 2 | 1
  Week 6: Indurated | 1 | 0
  Week 12: number analyzed (Participants) | 23 | 11
  Week 12: Normal | 21 | 8
  Week 12: Erythematous | 0 | 0
  Week 12: Edematous | 0 | 1
  Week 12: Eczematous | 0 | 1
  Week 12: Excoriated | 0 | 0
  Week 12: Macerated | 1 | 1
  Week 12: Indurated | 1 | 0

13. Secondary Outcome: Ulcer Progression Assessed by Change From Baseline in Wound Area
Description: The change from Baseline of the wound area was calculated to assess wound healing measured at each time point. Analyses were conducted using the last observation carried forward (LOCF) method to account for any missing follow-up visit data. A positive value indicated the wound showed an improvement in healing; a negative value indicated the wound showed worsening healing status based on wound area measurements.
Time Frame: Baseline, Weeks 3, 6 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
cm^2
  Baseline, wound area | 8.9 (11.9) | 8.7 (8.9)
  Week 3, wound area: number analyzed (Participants) | 24 | 11
  Week 3, wound area | 9.9 (13.3) | 4.9 (6.4)
  Week 3, change in wound area: number analyzed (Participants) | 24 | 11
  Week 3, change in wound area | -0.6 (10.6) | 2.2 (4.6)
  Week 6, wound area: number analyzed (Participants) | 24 | 11
  Week 6, wound area | 9.7 (16.1) | 3.7 (6.5)
  Week 6, change in wound area: number analyzed (Participants) | 24 | 11
  Week 6, change in wound area | -0.5 (12.2) | 3.3 (5.0)
  Week 12, wound area: number analyzed (Participants) | 24 | 12
  Week 12, wound area | 7.9 (15.8) | 6.7 (18.5)
  Week 12, change in wound area: number analyzed (Participants) | 24 | 12
  Week 12, change in wound area | 1.4 (13.7) | 0.0 (16.4)

14. Secondary Outcome: Ulcer Progression Assessed by Change From Baseline in Wound Volume
Description: The change from Baseline of the wound volume was calculated to assess wound healing measured at each time point. Analyses were conducted using the last observation carried forward (LOCF) method to account for any missing follow-up visit data. A positive value indicated the wound showed an improvement in healing; a negative value indicated the wound showed worsening healing status based on wound volume measurements.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
cm^3
  Baseline, wound volume | 2.7 (5.2) | 2.1 (2.6)
  Week 3, wound volume: number analyzed (Participants) | 24 | 11
  Week 3, wound volume | 2.5 (5.7) | 1.0 (1.9)
  Week 3, change in wound volume: number analyzed (Participants) | 24 | 11
  Week 3, change in wound volume | 0.3 (1.6) | 1.0 (1.7)
  Week 6, wound volume: number analyzed (Participants) | 24 | 11
  Week 6, wound volume | 2.9 (7.3) | 0.9 (2.6)
  Week 6, change in wound volume: number analyzed (Participants) | 24 | 11
  Week 6, change in wound volume | -0.1 (3.1) | 1.1 (2.3)
  Week 12, wound volume: number analyzed (Participants) | 24 | 12
  Week 12, wound volume | 2.2 (5.6) | 2.8 (9.3)
  Week 12, change in wound volume: number analyzed (Participants) | 24 | 12
  Week 12, change in wound volume | 0.6 (1.9) | -0.8 (8.0)

15. Secondary Outcome: Ulcer Progression Assessed by Change From Baseline in Wound Depth
Description: The change from Baseline in the wound depth was calculated to assess wound healing measured at each time point. Analyses were conducted using the last observation carried forward (LOCF) method to account for any missing follow-up visit data. A positive value indicated the wound showed an improvement in healing; a negative value indicated the wound showed worsening healing status based on wound depth measurements.
Time Frame: Baseline, Weeks 3, 6, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
mm
  Baseline, wound depth | 2.8 (3.6) | 3.8 (5.0)
  Week 3, wound depth: number analyzed (Participants) | 24 | 11
  Week 3, wound depth | 1.8 (1.8) | 2.7 (4.3)
  Week 3, change in wound depth: number analyzed (Participants) | 24 | 11
  Week 3, change in wound depth | 1.0 (2.9) | 1.2 (2.0)
  Week 6, wound depth: number analyzed (Participants) | 24 | 11
  Week 6, wound depth | 1.9 (2.3) | 1.5 (2.0)
  Week 6, change in wound depth: number analyzed (Participants) | 24 | 11
  Week 6, change in wound depth | 0.9 (3.3) | 2.4 (5.1)
  Week 12, wound depth: number analyzed (Participants) | 24 | 12
  Week 12, wound depth | 1.3 (1.9) | 0.9 (1.6)
  Week 12, change in wound depth: number analyzed (Participants) | 24 | 12
  Week 12, change in wound depth | 1.6 (3.7) | 3.1 (5.0)

16. Secondary Outcome: Number of Participants With Reference Wound Healed
Description: Assessment of the wound healed status (100% re-epithelialized, no drainage, no need for dressing) was analyzed at each visit to determine the healing status of the ulcer. Analyses were conducted using the last observation carried forward (LOCF) method to account for any missing follow-up visit data.
Time Frame: Weeks 3, 6 and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 24 | 13
Participants
  Week 3, reference ulcer healed: number analyzed (Participants) | 24 | 11
  Week 3, reference ulcer healed: No | 23 | 11
  Week 3, reference ulcer healed: Yes | 1 | 0
  Week 6, reference ulcer healed: number analyzed (Participants) | 24 | 11
  Week 6, reference ulcer healed: No | 22 | 10
  Week 6, reference ulcer healed: Yes | 2 | 1
  Week 12, reference ulcer healed: No | 15 | 8
  Week 12, reference ulcer healed: Yes | 9 | 5

17. Secondary Outcome: Healthcare Resource Use Related to the Reference Ulcer Over 12 Weeks - Number of Dressings Used
Description: Analysis of the healthcare resources used related to the reference ulcer included:
  Number of primary and secondary dressings including use of compression therapy.
Time Frame: Baseline through 12 weeks
Population: Two subjects in the standard care group withdrew prior to receiving treatment.
Measure: Mean (Standard Deviation); unit: dressings used/participant
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
dressings used/participant | 10.4 (4.8) | 18.3 (20.5)

18. Secondary Outcome: Healthcare Resource Use Related to the Reference Ulcer - Type of Dressings Used Per Dressing Change
Description: Analysis of the healthcare resources used related to the reference ulcer included:
  Type of primary and secondary dressings including compression therapy used during each dressing change over the 12-week treatment period based on the size of the ulcer.
Time Frame: Baseline through 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Dressings used per change
Units Other Than Participants: Dressings used per change
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Number analyzed (Dressings used per change) | 260 | 126
Dressings used per change
  ALLEVYN Life Non-bordered (ALNB), 10.5 x 10.5 cm: number analyzed (Participants) | 25 | 0
  ALLEVYN Life Non-bordered (ALNB), 10.5 x 10.5 cm: number analyzed (Dressings used per change) | 138 | 0
  ALLEVYN Life Non-bordered (ALNB), 10.5 x 10.5 cm | 1.0 (0.0) |
  ALNB, 16 x 16 cm: number analyzed (Participants) | 25 | 0
  ALNB, 16 x 16 cm: number analyzed (Dressings used per change) | 33 | 0
  ALNB, 16 x 16 cm | 1.0 (0.0) |
  ALNB, 10 x 20 cm: number analyzed (Participants) | 25 | 0
  ALNB, 10 x 20 cm: number analyzed (Dressings used per change) | 89 | 0
  ALNB, 10 x 20 cm | 1.0 (0.1) |
  Standard care: number analyzed (Participants) | 0 | 13
  Standard care: number analyzed (Dressings used per change) | 0 | 126
  Standard care |  | 1.9 (1.0)

19. Secondary Outcome: Healthcare Resource Use - Number and Type of Compression Dressings Used
Description: Not all enrolled participants required the use of compression dressings. Of those participants who did require a compression dressing, an analysis of the healthcare resources used included the number and type of primary and secondary dressings used in relation to the reference ulcer.
Time Frame: Baseline through 12 weeks
Population: Two subjects from the standard care group withdrew prior to receiving treatment.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Number analyzed (Wounds) | 68 | 33
Wounds
  Multi layer elastic - Profore | 16 | 7
  Multi layer elastic other than Profore | 15 | 8
  Multi layer inelastic | 0 | 0
  Single layer elastic | 2 | 2
  Single layer inelastic | 0 | 0
  Support hosiery | 0 | 1
  Other | 0 | 0
  Compression dressing application not required | 35 | 15

20. Secondary Outcome: Healthcare Resource Use - Number of Participants Requiring Hospital Admission
Description: Analysis of the healthcare resources used for participants who required a hospital admission related to the reference ulcer.
Time Frame: Baseline through 12 weeks
Population: Two subjects from the standard care group withdrew prior to receiving treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Participants | 0 | 1

21. Secondary Outcome: Healthcare Resource Use - Number of Days Participants Required In-Hospital Care
Description: Analysis of the healthcare resources used related to the reference ulcer included: Time in hospital (number of days spent as an inpatient due to reference ulcer).
Time Frame: Baseline through 12 weeks
Population: Two subjects from the standard care group withdrew prior to receiving treatment.
Measure: Number; unit: Days
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 0 | 1
Days |  | 7

22. Secondary Outcome: Healthcare Resource Use - Number of Dressing Changes Required for Each Type of Wound Debridement
Description: Analysis of the healthcare resources used related to the reference ulcer included:
  Interventions/procedures related to the reference ulcer (number and type) including debridement of the ulcer.
Time Frame: Baseline through 12 weeks
Population: Two subjects from the standard care group withdrew prior to receiving treatment.
Measure: Count of Units; unit: Dressing changes
Units Other Than Participants: Dressing changes
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
Number analyzed (Participants) | 25 | 13
Number analyzed (Dressing changes) | 264 | 126
Dressing changes
  Curette debridement | 33 | 11
  Scissors debridement | 0 | 0
  Scalpel debridement | 69 | 26
  Forceps debridement | 1 | 0
  Other type of debridement | 2 | 0
  Wound debridement not required as part of care | 159 | 89

ADVERSE EVENTS:
Time Frame: Baseline through 12 weeks of treatment/End of Study Visit.
Arm/Group | ALLEVYN Life Non-Bordered | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/25 | 3/15
Other Adverse Events (participants affected / at risk) | 3/25 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALLEVYN Life Non-Bordered (N=25) | Standard Care (N=15)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALLEVYN Life Non-Bordered (N=25) | Standard Care (N=15)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A possible limitation of this study might include the broad nature of the standard of care treatment arm; such as, varying from dressing types to antimicrobial therapy used to NPWT, which may have made a standardized comparison to the ALLEVYN Life Non-Bordered dressing difficult to assess thoroughly. Due to the nature of the physical differences in the dressings it was not possible to blind either subjects or the clinicians.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT03146845/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT03146845/SAP_001.pdf